CLINICAL TRIAL: NCT06145217
Title: Open-label, Non-randomized, Two-treatment, Single-period, Single Dose, Drug-drug Interaction Study to Evaluate the Effects of Omeprazole 40mg on the Pharmacokinetics of SPRYCEL® 100 mg Film-coated Tablets (Dasatinib) in Adult Human Subjects
Brief Title: An Drug-drug Interaction Study to Evaluate the Effects of Omeprazole 40mg on the Pharmacokinetics of SPRYCEL®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XS004-17
Record Dates: First submitted 2023-11-10; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Drug-drug Interaction Study
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Intervention Model Description: An open-label, non-randomized, two-treatment, single-period, single dose, drug-drug interaction study, which allows for independent establishment of the true intrasubject variability for dasatinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPRYCEL® (dasatinib) 100 mg Film-Coated Tablets (Experimental): To evaluate the drug-drug interaction between SPRYCEL® 100 mg (US sourced) and Omeprazole under fasted conditions in healthy, adult, human subjects.
  Interventions: Drug: SPRYCEL® (dasatinib) 100 mg Film-Coated Tablets in combination with Omeprazole Delayed-Release Capsules USP, 40 mg

INTERVENTIONS:
Drug: SPRYCEL® (dasatinib) 100 mg Film-Coated Tablets in combination with Omeprazole Delayed-Release Capsules USP, 40 mg — To evaluate the drug-drug interaction between SPRYCEL® 100 mg and Omeprazole under fasted conditions in healthy, adult, human subjects.
  Other Names: dasatinib

SUMMARY:
A drug-drug interaction study designed to evaluate the drug-drug interaction between SPRYCEL® 100 mg (US sourced) and Omeprazole in healthy, adult, human subjects

DETAILED DESCRIPTION:
A drug-drug interaction study and was designed to evaluate the drug-drug interaction between SPRYCEL® 100 mg (US sourced) and Omeprazole in healthy, adult, human subjects under fasted conditions at a time point when a high pH effect of omeprazole is expected, i.e., omeprazole at steady state and dasatinib are administered 9 hours apart. 18 healthy, adult, human subjects were enrolled into the study. Forty (40) PK blood sampling time points and a washout period of 05 days (between two administration of the study drug SPRYCEL® 100mg) were planned so that the drug concentration in the biological fluid could be characterized accurately for this drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human beings 18 and 45 years of age.
* Subjects weighing at least 50 kg for male or 45 kg for female, having a body mass index between 18.5 Kg/m2 and 29.9 Kg/m2.
* Subject must be able to provide written informed consent with a detailed description of nature of the drug.
* Acceptable medical history, physical examination, Electrocardiography (ECG), laboratory investigations within 21 days prior to enrollment and chest X-ray.
* Female subjects must meet one of the following criteria:

Physiological postmenopausal status, defined as the following. Absence of menses for at least one year prior to the first study drug administration (without an alternative medical condition); and FSH levels ≥40 mlU/mL during screening / at check-in or Surgical postmenopausal status. Must agree to use an adequate method of contraception. Bilateral tubal occlusion or hysterectomy

* Clinical laboratory values should be within the laboratory's stated normal range.
* The subject is able to communicate meaningfully with study personnel and is anticipated to be able to comply fully with study procedures
* Male or Female subjects who participate in the study should agree to practice abstention or contraception during the study and for at least 90 days after the last dose of dasatinib.
* Male subjects should not donate sperm for 90 days from the last administration of IMP.
* Light, Non or ex-smoker

Exclusion Criteria:

* Systolic blood pressure less than 100 mm of Hg or more than 140 mm of Hg.
* Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.
* Body temperature less than 95.0 °F (35.0 °C) or above 98.6°F (37.0 °C).
* Pulse rate less than 60/min or above 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.
* Any history of impairment of cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease, or disorder.
* History of hematological, bleeding, and malignant disorders
* History of gastrointestinal disorders that may affect the absorption of the drug, including achlorhydria, hypochlorhydria, hypermotility, hypomotility, malabsorption disorder, diarrhoea, prior bowel resection, colostomy, and ileostomy.
* Subjects with estimated glomerular filtration rate < 90 mL/minute/1.73 m2 at screening or on the day of check-in.
* History of taking anticoagulant medication, antiarrhythmics and antiplatelet agents.
* A prolonged QTc interval (QTc greater than 450 ms) demonstrated on ECG at Screening.
* Volunteer has taken P-gp inhibitors within 30 days prior to the check-in.
* History of any drug or alcohol abuse in the past 2 years.
* History of intake of strong CYP3A4 inhibitors (see Appendix-5) or inducers within 4 weeks prior to the check-in.
* History of intake of drugs known to prolong the QTc interval within 4 weeks prior to the check-in (see Appendix-5).
* Patients with rare hereditary problems of galactose intolerance, severe lactase deficiency with a severe degree of intolerance to lactose-containing products, or of glucose-galactose malabsorption.
* Any clinically significant ECG abnormalities that, in the Investigator's opinion, would compromise the subject's safety.
* Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
* History or family history of long QT syndrome.
* A history of difficulty with donating blood and having poor vein access.
* Male subjects with pregnant or lactating partners.
* Volunteers who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies, vitamins or minerals in the 14 days before check-in (other than up to 4 gr of paracetamol per day).
* Consumption of the xanthine containing food or beverages (like tea, coffee, chocolates, and flavored drinks) at least 48 hours before check-in.
* Consumption of the grapefruit or grapefruit juice, pomegranate, or pomegranate juice at least 14 days before check-in.
* Consumption of tobacco containing products (including smoking cigarettes or chewing tobacco products), e-cigarettes and/or nicotine replacement products within 3 months prior to the check-in.
* Consumption of all kinds of alcoholic beverages from at least 48.00 hours prior to check-in until the last blood sample collection in study period.
* Difficulty in abstaining from all kinds of alcoholic beverages during entire study period.
* Difficulty in abstaining from the xanthine containing food or beverages (like tea, coffee, chocolates, and flavored drinks), grapefruit or grapefruit juice, pomelo, pomegranate, or pomegranate juice during entire study period.
* Difficulty in abstaining from the smoking or chewing tobacco products during entire study period.
* Intake of any medication in last 30 days except caffeine, ranitidine, paracetamol, diclofenac sodium and ondansetron.
* Confirmed positive drugs of abuse (benzodiazepines, tetrahydrocannabinol, amphetamine, cocaine, barbiturates, and morphine) on check-in.
* Confirmed positive alcohol (breath) test on check-in.
* Confirmed positive Covid-19 Rapid Antigen test on check-in.
* Participated in any other clinical study or donated blood in last 90 days.
* Intake of pomelo, starfruit, Seville oranges, and St. John's Wort within the previous 14 days before check-in.
* Difficulty in abstaining from the pomelo, starfruit, Seville oranges, and St. John's Wort throughout the study.
* Positive screens for serum hepatitis B surface antigen (HbsAg), hepatitis C antibody (HepC) or human immunodeficiency virus (HIV).
* Participated in contact sports or unaccustomed strenuous exercise in the 72 hours before check-in of any period.
* History of clinically significant allergy.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* History of allergy or sensitivity to dasatinib, or history of any food or drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* History of chronic infectious disease, system disorders, organ dysfunction especially cardiovascular disorders (e.g., arterial vascular occlusive events), respiratory disorders, renal or hepatic disorders, diabetes, or obesity.
* Volunteers having greater than the upper limit of normal values of Alkaline phosphatase (ALP), alanine transaminase (ALT), aspartate aminotransferase (AST) and total bilirubin.
* Clinically significant hypokalemia, hypomagnesemia, or other electrolyte disorders.
* Volunteers with history of malignant disorders.
* Volunteers with history of hematological, bleeding disorders.
* Volunteers on anticoagulant therapy.
* History of gastrointestinal disease or history of malabsorption within the last year, as determined by the Investigator.
* Confirmed positive pregnancy test (for females) on check-in.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Drug-drug interaction Plasma Concentration (Cmax) | a time point when a high potential hydrogen (pH) effect of omeprazole is expected, i.e., omeprazole at steady state and dasatinib are administered 9 hours apart.
  To evaluate the drug-drug interaction between SPRYCEL® 100 mg and Omeprazole in healthy, adult, human subjects under fasted conditions at a time point when a high pH effect of omeprazole is expected. Dasatinib (SPRYCEL®) concentration-time profiles will be evaluated using non-compartmental methods. Peak Plasma Concentration (Cmax) and tmax will be derived from the observed plasma concentration data.
Drug-drug interaction AUC0-t | a time point when a high potential hydrogen (pH) effect of omeprazole is expected, i.e., omeprazole at steady state and dasatinib are administered 9 hours apart.
  To evaluate the drug-drug interaction between SPRYCEL® 100 mg and Omeprazole in healthy, adult, human subjects under fasted conditions at a time point when a high pH effect of omeprazole is expected. Dasatinib (SPRYCEL®) concentration-time profiles will be evaluated using non-compartmental methods. AUC0-t will be calculated using linear trapezoidal interpolation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, Study Director — Xspray Pharma AB
Locations (1):
- QPS Bioserve India Pvt Limited, Hyderabad, India

IPD SHARING:
Plan to Share IPD: No